CLINICAL TRIAL: NCT02471911
Title: A Phase I Investigator-Initiated Study of Selinexor (KPT-330) Plus RICE in Patients With Relapsed or Refractory Aggressive B-cell Lymphomas
Brief Title: KPT-330 Plus RICE for Relapsed/Refractory Aggressive B-Cell Lymphoma
Acronym: KPT-330+RICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); The Leukemia and Lymphoma Society (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1502015891
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; Aggressive; Diffuse; Large
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Aggression | interventions — selinexor; Rituximab; Etoposide; Carboplatin; Ifosfamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects will receive KPT-330 (selinexor) on days -5 and -3 starting one week before RICE chemotherapy is started. Once chemotherapy starts, selinexor will be given on days 1, 3, and 5 of each chemotherapy cycle.
  RICE chemotherapy will consist of Rituximab, ifosfamide, carboplatin, etoposide, and dexamethasone.
  Interventions: Drug: KPT-330; Drug: Rituximab; Drug: Etoposide; Drug: Carboplatin; Drug: Ifosfamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: KPT-330 — KPT-330 administered orally on days -5 and -3 prior to starting chemotherapy. Once chemotherapy starts, KPT-330 will be administered on days 1, 3, and 5 of each cycle. Dose levels will range from 20 mg to 100mg with a standard 3+3 escalation schema.
  Other Names: Selinexor
Drug: Rituximab — IV Rituximab 375 mg/m2 on D1
  Other Names: Rituxan
Drug: Etoposide — IV Etoposide 100 mg/m2 on D1-3
Drug: Carboplatin — IV Carboplatin AUC 5 on D2
Drug: Ifosfamide — IV Ifosfamide 5 g/m2 on D2
Drug: Dexamethasone — 20 mg qd on Days -5 and -3. 20 mg qd on Days 1-5

SUMMARY:
This study evaluates the addition of selinexor (KPT-330) to RICE chemotherapy in the treatment of relapsed and refractory aggressive B-Cell Lymphoma, with the goal of improved response rates (as compared to RICE chemotherapy alone).

DETAILED DESCRIPTION:
Although aggressive B-cell lymphomas are potentially curable with front-line chemotherapy, at least one-third of patients experience progression or relapse. Second-line regimens such as rituximab, ifosfamide, carboplatin, and etoposide (RICE) are administered with the goal of cytoreduction prior to autologous stem cell transplantation (ASCT) in eligible patients. However, half of patients who receive salvage treatment and ASCT are still not cured.

Selinexor is a Selective Inhibitor of Nuclear Export / SINE compound, which is a new class of molecule. SINE compounds have been shown to induce apoptotic cell death in pre-clinical models of AML, CLL, T-ALL, and Ph+ ALL as well as B and T-cell non-Hodgkin lymphomas. Preliminarily, selinexor has demonstrated promising single-agent clinical activity in patients with previously treated NHL including DLBCL, warranting further investigation. Based on promising preclinical and clinical data, selinexor is currently under evaluation in combination with chemotherapy for solid tumors.

The investigators hypothesize that the combination of selinexor plus RICE will be well-tolerated and clinically active in participants with previously treated aggressive B-cell lymphomas and propose a phase I trial to evaluate this combination. Moreover, Investigators will evaluate primary patient samples before and after selinexor to investigate the mechanisms of action of selinexor, including the mechanisms by which selinexor sensitizes cells to chemotherapy, and evaluate other novel drug combinations in aggressive B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed aggressive B-cell non-Hodgkin lymphomas:

  * DLBCL including ABC, GCB or PMBCL subtypes
  * Double/triple hit lymphomas
  * Indolent lymphomas transformed to aggressive lymphomas
  * Follicular lymphomas grade 3B
* Patients must have received at least two cycles of anthracycline based chemotherapy administered with curative intent and one of the following:

  * failed to have achieve at least a partial response after 2 or more cycles
  * failed to achieve a complete response after 6 or more cycles
  * progressed after an initial response
* Patients must be age ≥18 years.
* Patients must have at least one site of measurable disease, 1.5 cm in diameter or greater.
* Patients must have ECOG performance status of 0-2.
* Patients must have laboratory test results within these ranges:

  * Absolute neutrophil count ≥ 1500/mm³
  * Platelet count ≥ 100,000/mm³
  * Serum creatinine clearance ≥40 mL/min
  * Total bilirubin ≤ 1.5x ULN. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
  * AST (SGOT) and ALT (SGPT) ≤ 2x ULN
* Women of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test prior to selinexor treatment. Male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential.

  * Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal.
  * For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Patients must be able to understand and willing to sign a written informed consent document.
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patients must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

Exclusion Criteria:

* Patients with hyperuricemia or other potential signs of tumor lysis syndrome
* Patients with more than minimally symptomatic disease (i.e. > grade 1), high tumor burden, or other indication for urgent treatment.
* Patients who have had prior malignancies (other than B-cell lymphomas) for ≤5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Patients who have had other anti-cancer therapy, including radiation or experimental drug or therapy, within 28 days of enrollment.
* Patients with known HIV, active hepatitis B, active hepatitis C.
* Patients with known central nervous system involvement by lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dosage (MTD) of Selinexor/KPT-330 when combined with RICE chemo in a relapsed/refractory aggressive b-cell lymphoma setting. | approximately 24 months
  The highest dose level at which no more than 1 or 6 patients presents with a dose-limiting toxicity (DLT) during the first 6 cycles of treatment

SECONDARY OUTCOMES:
Survival of subjects treated with KPT-330 + RICE | approximately 24 months per patient
  Overall survival of patients enrolled on KPT-330 + RICE
Progression-Free Survival of subjects treated with KPT-330 + RICE | approximately 24 months per patient
  Progression-free survival of patients enrolled on KPT-330+RICE
Number of patients who demonstrate a Response to KPT-330+RICE | approximately 24 months per patient
  The efficacy (as assessed by clinical response) of the combination of KPT-330 + RICE in patients with Rel/Ref b-cell lymphoma
Number of patients who undergo stem cell collection after induction therapy with KPT-330 + RICE | approximately 24 months per patient
  The number of patients who can feasibly undergo a stem cell transplant after treatment with KPT-330+RICE

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States